CLINICAL TRIAL: NCT01200056
Title: A Prospective, Double-blinded, Randomised Study to Evaluate the Effects of Different Doses of Statin Treatment on Plaque Volume and Composition in Coronary Disease Determined by Virtual Histology Using Intravascular Ultrasound
Brief Title: Virtual Histology Findings and Effects of Varying Doses of Atorvastatin Treatment
Acronym: VENUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prof. Stephen Lee (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Prof. Stephen Lee, Professor and Chief, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW 07-266 (IRB HKU); HKCTR-517 (Other: Clinical Trials Centre, HKU (www.HKClinicalTrials.com))
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Coronary Disease; Ultrasonography, Interventional; Hydroxymethylglutaryl-CoA Reductase Inhibitors
Keywords: Volumetric virtual histology intravascular ultrasound.; Statin-naive patient.; Varying doses atorvastatin.; Clinical outcomes.
MeSH Terms: conditions — Coronary Disease | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin 10mg low dose (Active Comparator): Atorvastatin 10mg daily for 6 months and compared to atorvastatin 40mg daily in the other arm. The primary endpoint of 6 months VH-IVUS findings and clinical outcomes would be monitored and compared.
  Interventions: Drug: Atorvastatin 10mg versus 40mg.
- Atorvastatin 40mg moderate dose (Active Comparator): Atorvastatin 40mg daily for 6 months and compared to atorvastatin 10mg daily in the other arm. The primary endpoint of 6 months VH-IVUS findings and clinical outcomes would be monitored and compared.
  Interventions: Drug: Atorvastatin 10mg versus 40mg.

INTERVENTIONS:
Drug: Atorvastatin 10mg versus 40mg. — 2 arms comparing atorvastatin 10mg daily for 6 months to atorvastatin 40mg daily for 6 months. The primary endpoint would be the 6 months VH-IVUS findings and clinical outcomes.
  Other Names: Lipitor 10mg versus 40mg daily for 6 months.

SUMMARY:
While statin treatment may induce plaque regression, the effect of statin on plaque composition with varying doses is unknown. This study assessed such effects by volumetric virtual histology intravascular ultrasound (VH-IVUS).

In this prospective, randomized, double-blinded pilot study, statin-naïve patients with stable angina requiring percutaneous coronary intervention (PCI) were randomized to receive 6 months of either atorvastatin 10mg or 40 mg daily. VH-IVUS was performed in all non-PCI lesions at baseline and 6 months; all analyses were performed by core laboratory.

DETAILED DESCRIPTION:
Statin therapy, especially at intensive doses, is beneficial in atherosclerotic coronary disease. Detecting subtle plaque regression after statin therapy is difficult by coronary angiogram; intravascular ultrasound (IVUS) is a far better method. Volumetric IVUS has been used in statin trials to evaluate plaque regression. Intensive statin therapy in the REVERSAL Trial and ASTEROID Trial appeared to achieve better regression outcomes. Stable fibrous plaque is likely to be responsible for stable ischemia, while unstable plaque (large lipid core, calcified nodule and necrotic core), thin-cap fibroatheroma, plaque erosion and plaque rupture may be responsible for acute coronary syndrome (ACS). In vivo tissue characterization of plaque composition is therefore important, yet in this regard grayscale IVUS is insufficient. The development of Virtual Histology (VH) utilizing IVUS generated radiofrequency backscattering signals to virtually separate plaque composition into 4 components corresponding to histopathology has made possible in vivo assessment of plaque composition and stability. We believed plaque regression and VH-IVUS plaque modification with statin therapy could be statin dose dependent, and may affect clinical outcomes. This study was designed to prove our hypothesis, utilizing VH-IVUS.

This study is the first prospective, randomised, double-blinded pilot study designed to investigate the varying statin dose effects on plaque regression and VH composition modulation. For ethical reasons, a placebo arm was not designed. Based on available data, clinically realistic doses of atorvastatin 10mg (low dose) and 40mg (moderate dose) were chosen. Only statin-naïve patients without previous history of myocardial infarction (MI) would be selected, aiming to show the "pure" effects of varying doses of statin and to better reveal the subtle differences in the changes.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 85 (not pregnant) requiring percutaneous intervention to coronary stenosis.
* Statin naive patient.
* No history of myocardial infarction. Angina free for at least 8 weeks.

Exclusion Criteria:

* Any history of previous statin treatment and myocardial infarction
* Current acute coronary syndrome or in cardiogenic shock
* Surgical bypass candidate
* Chronic total occlusion and very tortuous calcified arteries precluding safe IVUS examination.
* Patient refused to give written informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-08; Primary Completion 2009-11 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint would be the 6-month angiographic and VH-IVUS restudy findings. | 6 months
  Our hypothesis was plaque regression and virtual histology intravascular ultrasound (VH-IVUS) plaque modification with statin therapy could be statin dose dependent, and may affect clinical outcomes. 2 clinically realistic doses of atorvastatin 10mg and 40mg were chosen in statin-naïve patients without previous myocardial infarction. The primary endpoint of this study would therefore be the 6 months angiographic and IVUS follow-up, looking at the volumetric gray-scale IVUS and VH-IVUS findings at 6 months for the whole cohort as well as the differences between the 2 groups.

SECONDARY OUTCOMES:
The secondary endpoint would be the occurrence of any major adverse cardiac events at 6 months (including any death, myocardial infarction or need for revascularization) as routinely monitored after all percutaneous interventional procedures. | Throughout the 6 months study period.
  As described in the "Title" above.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Stephen WL LEE, MD FRCP FACC, Principal Investigator — Department of Medicine, the University of Hong Kong, Queen Mary Hospital, Hospital Authority
Locations (1):
- Department of Medicine, the University of Hong Kong, Queen Mary Hospital, Hospital Authority, Hong Kong SAR, Hong Kong, China

REFERENCES:
- [Background] Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults. Executive Summary of The Third Report of The National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, And Treatment of High Blood Cholesterol In Adults (Adult Treatment Panel III). JAMA. 2001 May 16;285(19):2486-97. doi: 10.1001/jama.285.19.2486. No abstract available. PMID 11368702
- [Background] De Backer G, Ambrosioni E, Borch-Johnsen K, Brotons C, Cifkova R, Dallongeville J, Ebrahim S, Faergeman O, Graham I, Mancia G, Manger Cats V, Orth-Gomer K, Perk J, Pyorala K, Rodicio JL, Sans S, Sansoy V, Sechtem U, Silber S, Thomsen T, Wood D; Third Joint Task Force of European and Other Societies on Cardiovascular Disease Prevention in Clinical Practice. European guidelines on cardiovascular disease prevention in clinical practice. Third Joint Task Force of European and Other Societies on Cardiovascular Disease Prevention in Clinical Practice. Eur Heart J. 2003 Sep;24(17):1601-10. doi: 10.1016/s0195-668x(03)00347-6. No abstract available. PMID 12964575
- [Background] Heart Protection Study Collaborative Group. MRC/BHF Heart Protection Study of cholesterol lowering with simvastatin in 20,536 high-risk individuals: a randomised placebo-controlled trial. Lancet. 2002 Jul 6;360(9326):7-22. doi: 10.1016/S0140-6736(02)09327-3. PMID 12114036
- [Background] Grundy SM, Cleeman JI, Merz CN, Brewer HB Jr, Clark LT, Hunninghake DB, Pasternak RC, Smith SC Jr, Stone NJ; National Heart, Lung, and Blood Institute; American College of Cardiology Foundation; American Heart Association. Implications of recent clinical trials for the National Cholesterol Education Program Adult Treatment Panel III guidelines. Circulation. 2004 Jul 13;110(2):227-39. doi: 10.1161/01.CIR.0000133317.49796.0E. PMID 15249516
- [Background] Schwartz GG, Olsson AG, Ezekowitz MD, Ganz P, Oliver MF, Waters D, Zeiher A, Chaitman BR, Leslie S, Stern T; Myocardial Ischemia Reduction with Aggressive Cholesterol Lowering (MIRACL) Study Investigators. Effects of atorvastatin on early recurrent ischemic events in acute coronary syndromes: the MIRACL study: a randomized controlled trial. JAMA. 2001 Apr 4;285(13):1711-8. doi: 10.1001/jama.285.13.1711. PMID 11277825
- [Background] Koren MJ, Hunninghake DB; ALLIANCE Investigators. Clinical outcomes in managed-care patients with coronary heart disease treated aggressively in lipid-lowering disease management clinics: the alliance study. J Am Coll Cardiol. 2004 Nov 2;44(9):1772-9. doi: 10.1016/j.jacc.2004.07.053. PMID 15519006
- [Background] LaRosa JC, Grundy SM, Waters DD, Shear C, Barter P, Fruchart JC, Gotto AM, Greten H, Kastelein JJ, Shepherd J, Wenger NK; Treating to New Targets (TNT) Investigators. Intensive lipid lowering with atorvastatin in patients with stable coronary disease. N Engl J Med. 2005 Apr 7;352(14):1425-35. doi: 10.1056/NEJMoa050461. Epub 2005 Mar 8. PMID 15755765
- [Background] Cannon CP, Braunwald E, McCabe CH, Rader DJ, Rouleau JL, Belder R, Joyal SV, Hill KA, Pfeffer MA, Skene AM; Pravastatin or Atorvastatin Evaluation and Infection Therapy-Thrombolysis in Myocardial Infarction 22 Investigators. Intensive versus moderate lipid lowering with statins after acute coronary syndromes. N Engl J Med. 2004 Apr 8;350(15):1495-504. doi: 10.1056/NEJMoa040583. Epub 2004 Mar 8. PMID 15007110
- [Background] Brown G, Albers JJ, Fisher LD, Schaefer SM, Lin JT, Kaplan C, Zhao XQ, Bisson BD, Fitzpatrick VF, Dodge HT. Regression of coronary artery disease as a result of intensive lipid-lowering therapy in men with high levels of apolipoprotein B. N Engl J Med. 1990 Nov 8;323(19):1289-98. doi: 10.1056/NEJM199011083231901. PMID 2215615
- [Background] Hausmann D, Erbel R, Alibelli-Chemarin MJ, Boksch W, Caracciolo E, Cohn JM, Culp SC, Daniel WG, De Scheerder I, DiMario C, et al. The safety of intracoronary ultrasound. A multicenter survey of 2207 examinations. Circulation. 1995 Feb 1;91(3):623-30. doi: 10.1161/01.cir.91.3.623. PMID 7828285
- [Background] Potkin BN, Bartorelli AL, Gessert JM, Neville RF, Almagor Y, Roberts WC, Leon MB. Coronary artery imaging with intravascular high-frequency ultrasound. Circulation. 1990 May;81(5):1575-85. doi: 10.1161/01.cir.81.5.1575. PMID 2184946
- [Background] Tobis JM, Mallery J, Mahon D, Lehmann K, Zalesky P, Griffith J, Gessert J, Moriuchi M, McRae M, Dwyer ML, et al. Intravascular ultrasound imaging of human coronary arteries in vivo. Analysis of tissue characterizations with comparison to in vitro histological specimens. Circulation. 1991 Mar;83(3):913-26. doi: 10.1161/01.cir.83.3.913. PMID 1999040
- [Background] Mintz GS, Nissen SE, Anderson WD, Bailey SR, Erbel R, Fitzgerald PJ, Pinto FJ, Rosenfield K, Siegel RJ, Tuzcu EM, Yock PG. American College of Cardiology Clinical Expert Consensus Document on Standards for Acquisition, Measurement and Reporting of Intravascular Ultrasound Studies (IVUS). A report of the American College of Cardiology Task Force on Clinical Expert Consensus Documents. J Am Coll Cardiol. 2001 Apr;37(5):1478-92. doi: 10.1016/s0735-1097(01)01175-5. No abstract available. PMID 11300468
- [Background] Mintz GS, Painter JA, Pichard AD, Kent KM, Satler LF, Popma JJ, Chuang YC, Bucher TA, Sokolowicz LE, Leon MB. Atherosclerosis in angiographically "normal" coronary artery reference segments: an intravascular ultrasound study with clinical correlations. J Am Coll Cardiol. 1995 Jun;25(7):1479-85. doi: 10.1016/0735-1097(95)00088-l. PMID 7759694
- [Background] Nissen SE, Tuzcu EM, Schoenhagen P, Brown BG, Ganz P, Vogel RA, Crowe T, Howard G, Cooper CJ, Brodie B, Grines CL, DeMaria AN; REVERSAL Investigators. Effect of intensive compared with moderate lipid-lowering therapy on progression of coronary atherosclerosis: a randomized controlled trial. JAMA. 2004 Mar 3;291(9):1071-80. doi: 10.1001/jama.291.9.1071. PMID 14996776
- [Background] Nissen SE. Application of intravascular ultrasound to characterize coronary artery disease and assess the progression or regression of atherosclerosis. Am J Cardiol. 2002 Feb 21;89(4A):24B-31B. doi: 10.1016/s0002-9149(02)02217-8. PMID 11879665
- [Background] Takagi T, Yoshida K, Akasaka T, Hozumi T, Morioka S, Yoshikawa J. Intravascular ultrasound analysis of reduction in progression of coronary narrowing by treatment with pravastatin. Am J Cardiol. 1997 Jun 15;79(12):1673-6. doi: 10.1016/s0002-9149(97)00221-x. PMID 9202362
- [Background] Schartl M, Bocksch W, Koschyk DH, Voelker W, Karsch KR, Kreuzer J, Hausmann D, Beckmann S, Gross M. Use of intravascular ultrasound to compare effects of different strategies of lipid-lowering therapy on plaque volume and composition in patients with coronary artery disease. Circulation. 2001 Jul 24;104(4):387-92. doi: 10.1161/hc2901.093188. PMID 11468198
- [Background] Jensen LO, Thayssen P, Pedersen KE, Stender S, Haghfelt T. Regression of coronary atherosclerosis by simvastatin: a serial intravascular ultrasound study. Circulation. 2004 Jul 20;110(3):265-70. doi: 10.1161/01.CIR.0000135215.75876.41. Epub 2004 Jul 6. PMID 15238460
- [Background] Okazaki S, Yokoyama T, Miyauchi K, Shimada K, Kurata T, Sato H, Daida H. Early statin treatment in patients with acute coronary syndrome: demonstration of the beneficial effect on atherosclerotic lesions by serial volumetric intravascular ultrasound analysis during half a year after coronary event: the ESTABLISH Study. Circulation. 2004 Aug 31;110(9):1061-8. doi: 10.1161/01.CIR.0000140261.58966.A4. Epub 2004 Aug 23. PMID 15326073
- [Background] Kimura BJ, Bhargava V, DeMaria AN. Value and limitations of intravascular ultrasound imaging in characterizing coronary atherosclerotic plaque. Am Heart J. 1995 Aug;130(2):386-96. doi: 10.1016/0002-8703(95)90457-3. PMID 7631624
- [Background] Moore MP, Spencer T, Salter DM, Kearney PP, Shaw TR, Starkey IR, Fitzgerald PJ, Erbel R, Lange A, McDicken NW, Sutherland GR, Fox KA. Characterisation of coronary atherosclerotic morphology by spectral analysis of radiofrequency signal: in vitro intravascular ultrasound study with histological and radiological validation. Heart. 1998 May;79(5):459-67. doi: 10.1136/hrt.79.5.459. PMID 9659192
- [Background] Watson RJ, McLean CC, Moore MP, Spencer T, Salter DM, Anderson T, Fox KA, McDicken WN. Classification of arterial plaque by spectral analysis of in vitro radio frequency intravascular ultrasound data. Ultrasound Med Biol. 2000 Jan;26(1):73-80. doi: 10.1016/s0301-5629(99)00112-x. PMID 10687795
- [Background] Nair A, Kuban BD, Tuzcu EM, Schoenhagen P, Nissen SE, Vince DG. Coronary plaque classification with intravascular ultrasound radiofrequency data analysis. Circulation. 2002 Oct 22;106(17):2200-6. doi: 10.1161/01.cir.0000035654.18341.5e. PMID 12390948
- [Background] Nasu K, Tsuchikane E, Katoh O, Vince DG, Virmani R, Surmely JF, Murata A, Takeda Y, Ito T, Ehara M, Matsubara T, Terashima M, Suzuki T. Accuracy of in vivo coronary plaque morphology assessment: a validation study of in vivo virtual histology compared with in vitro histopathology. J Am Coll Cardiol. 2006 Jun 20;47(12):2405-12. doi: 10.1016/j.jacc.2006.02.044. Epub 2006 May 30. PMID 16781367
- [Background] Rodriguez-Granillo GA, Garcia-Garcia HM, Mc Fadden EP, Valgimigli M, Aoki J, de Feyter P, Serruys PW. In vivo intravascular ultrasound-derived thin-cap fibroatheroma detection using ultrasound radiofrequency data analysis. J Am Coll Cardiol. 2005 Dec 6;46(11):2038-42. doi: 10.1016/j.jacc.2005.07.064. Epub 2005 Nov 9. PMID 16325038
- [Background] Kolodgie FD, Burke AP, Farb A, Gold HK, Yuan J, Narula J, Finn AV, Virmani R. The thin-cap fibroatheroma: a type of vulnerable plaque: the major precursor lesion to acute coronary syndromes. Curr Opin Cardiol. 2001 Sep;16(5):285-92. doi: 10.1097/00001573-200109000-00006. PMID 11584167
- [Background] Virmani R, Burke AP, Kolodgie FD, Farb A. Vulnerable plaque: the pathology of unstable coronary lesions. J Interv Cardiol. 2002 Dec;15(6):439-46. doi: 10.1111/j.1540-8183.2002.tb01087.x. PMID 12476646
- [Background] Rioufol G, Finet G, Ginon I, Andre-Fouet X, Rossi R, Vialle E, Desjoyaux E, Convert G, Huret JF, Tabib A. Multiple atherosclerotic plaque rupture in acute coronary syndrome: a three-vessel intravascular ultrasound study. Circulation. 2002 Aug 13;106(7):804-8. doi: 10.1161/01.cir.0000025609.13806.31. PMID 12176951 (Retraction: PMID 22689939 Circulation. 2012 Jun 12;125(23):e1019)
- [Background] Rioufol G, Gilard M, Finet G, Ginon I, Boschat J, Andre-Fouet X. Evolution of spontaneous atherosclerotic plaque rupture with medical therapy: long-term follow-up with intravascular ultrasound. Circulation. 2004 Nov 2;110(18):2875-80. doi: 10.1161/01.CIR.0000146337.05073.22. Epub 2004 Oct 18. PMID 15492303
- [Background] Steinberg D. Thematic review series: the pathogenesis of atherosclerosis. An interpretive history of the cholesterol controversy: part II: the early evidence linking hypercholesterolemia to coronary disease in humans. J Lipid Res. 2005 Feb;46(2):179-90. doi: 10.1194/jlr.R400012-JLR200. Epub 2004 Nov 16. PMID 15547293